CLINICAL TRIAL: NCT00617643
Title: Comparison of Nevirapine Levels With and Without Dose Escalation in HIV-infected Patients Commencing Antiretroviral Therapy Who Are Also Receiving Rifampicin Based Anti-tuberculous Therapy
Brief Title: Nevirapine Drug Levels in HIV Positive Patients Also Receiving Rifampicin for Tuberculosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Liverpool (Other)
Responsible Party: Dr. Concepta Merry, Infectious Diseases Institute, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPR 004
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Nevirapine; Rifampicin; Pharmacokinetics
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Triomune® 30 one tablet once daily (am) plus Zerit® 30 + Epivir 150mg once daily (pm) for two weeks
  Interventions: Drug: Nevirapine initiation with dose escalation
- 1 (Experimental): Triomune® 30 one tablet twice daily for two weeks
  Interventions: Drug: Nevirapine without dose escalation

INTERVENTIONS:
Drug: Nevirapine without dose escalation — Fixed dose combination tablets of stavudine 30mg,lamivudine 150mg and nevirapine tablets 200mg twice daily at initiation of antiretroviral therapy in patients receiving rifampicin for tuberculosis therapy
  Other Names: Triomune 30
  Arms: 1
Drug: Nevirapine initiation with dose escalation — Triomune® 30 (according to body weight) one tablet once daily (am) plus Zerit® 30 + Epivir 150mg once daily (pm) for two weeks
  Arms: 2

SUMMARY:
Triomune is the most commonly prescribed treatment for HIV infection in Uganda. Triomune is manufactured by a generic drug company and consists of three drugs combined in a single pill given twice daily (stavudine 30mg plus lamivudine 150mg plus nevirapine 200mg).

It is known that the levels of nevirapine in a patient's blood are highest in the first two weeks of treatment. Therefore it is recommended that patients starting on nevirapine should undergo dose escalation i.e start on 200mg once daily for two weeks and then increase to full dose of 200mg twice daily in order to avoid nevirapine related rash. It is not possible to do dose escalation with a fixed dose combination pill like Triomune and for the two weeks of the dose escalation patients either can buy stavudine plus lamivudine plus nevirapine as separate pills or take Triomune in the morning and then take stavudine plus lamivudine as separate pills in the evening.

Rifampicin is used to treat TB and lowers the levels of nevirapine in a patient's blood. This raises two questions in routine clinical practice for patients who are co-infected with HIV and TB (1) Do we need to put our patients to the trouble of dose escalation of nevirapine if they are already on rifampicin? and (2) If we dose escalate nevirapine in patients on rifampicin, are we putting them at risk of low drug levels and development of resistance? The aim of this study is to compare the plasma concentrations of nevirapine in HIV infected patients who are commencing antiretroviral therapy with and without a lead in dose of nevirapine and who are also receiving concomitant treatment with antituberculous therapy which includes rifampicin to assess whether dose escalation of nevirapine is appropriate in this patient population

DETAILED DESCRIPTION:
Many patients in Uganda are co-infected with HIV and TB and require simultaneous treatment for both diseases. There is a paucity of data on the complex pharmacokinetic interactions between antiretroviral and anti-TB drugs and the available data is not representative of the African setting, hence it is important that these complex drug interactions be characterized fully.

Rifampicin is a potent inducer of several liver and intestinal enzymes responsible for drug metabolism including the cytochrome P450 (CYP450) system, and p-glycoprotein (PgP, a multi-drug resistant transport protein). The non-nucleoside reverse transcriptase inhibitors (NNRTIs) such as nevirapine are lipophilic drugs which undergo passive diffusion through the gastrointestinal lining. Once inside intestinal cells these drugs can be transported back to the luminal surface by PgP or oxidatively metabolised by CYP450 enzymes. Thus induction of CYP450 and PgP by rifampicin results in accelerated and more extensive presystemic metabolism of the NNRTI substrates resulting in decreased oral bioavailability. Available data suggests that rifampicin reduces the AUC of the NNRTI, nevirapine by 31% and the Cmin by 21% to 68% (Ribera 2001, Robinson 1998) respectively. While minor reductions in levels of the nucleoside reverse transcriptase inhibitor (NRTI), zidovudine have been reported (probably due to increased glucuronidation; (Burger 1993), it is generally agreed that the efficacy of the NRTIs is not affected by concomitant rifampicin use.

Nevirapine, a dipyridodiazepinone, is an inducer of cytochrome P450 and also induces its own metabolism with a reduction in the elimination half life from 45 to 25 hours on repeat dosing (Havlir, Murphy). The recommended daily dosing regimen of nevirapine for adults is 200mg twice daily. This is preceded by a two week lead in dose of 200mg once daily because of the autoinduction of nevirapine hepatic metabolism. This dose escalation strategy reduced nevirapine related rash from 48% (in the absence of dose escalation) to 18 %.( Murphy). Dose escalation of nevirapine is complex in the resource limited setting where fixed dose combinations of generically manufactured drugs are commonly prescribed. It is unclear as to whether dose escalation of nevirapine is necessary in patients on rifampicin as they already have full induction of their cytochrome P450 system provided that they have been on rifampicin for a minimum of two weeks. Furthermore, there is concern that dose escalation of nevirapine in this group of patients may expose patients to sub-therapeutic levels of nevirapine with the attendant risk of development of drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide full informed written consent
* Confirmed diagnosis of HIV infection
* On rifampicin therapy for at least two weeks
* Clinical criteria for commencing antiretroviral therapy

Exclusion Criteria:

* Hemoglobin < 8g/dl
* Liver and renal function tests > 3 times the upper limit of normal
* Pregnancy
* Use of know inhibitors or inducers of Cytochrome P450 or P-glycoprotein.
* Use of herbal medications
* Intercurrent Illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacokinetics of nevirapine with dose escalation and without dose escalation of nevirapine on day 7, 14 and 21 in patients who are on rifampicin therapy. | 12 months

SECONDARY OUTCOMES:
Safety and tolerability of nevirapine when administered in HIV-TB coinfected patients receiving rifampicin | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Concepta A Merry, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Infectious Diseases Institute, Faculty of Medicine, Makerere University, Kampala, Uganda

REFERENCES:
- [Derived] Lamorde M, Byakika-Kibwika P, Okaba-Kayom V, Ryan M, Coakley P, Boffito M, Namakula R, Kalemeera F, Colebunders R, Back D, Khoo S, Merry C. Nevirapine pharmacokinetics when initiated at 200 mg or 400 mg daily in HIV-1 and tuberculosis co-infected Ugandan adults on rifampicin. J Antimicrob Chemother. 2011 Jan;66(1):180-3. doi: 10.1093/jac/dkq411. Epub 2010 Nov 2. PMID 21047828